CLINICAL TRIAL: NCT02688647
Title: A Randomized, Phase 2, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability, and Activity of Belumosudil in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A 2-Part, Phase 2 Open-label and Crossover Study of Belumosudil for Treatment of Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KD025-207
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Results first posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Pulmonary Fibrosis; Fibrosis; Idiopathic Interstitial Pneumonias; Lung Diseases
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Fibrosis; Idiopathic Interstitial Pneumonias; Lung Diseases | interventions — belumosudil; KD025

STUDY DESIGN:
Intervention Model Description: In Part 1: Subjects are randomized to treatment with either Belumosudil 400 mg PO QD (Belumosudil-R) or to BSC (BSC-R).
  In Part 2: Subjects who are randomized and receive Belumosudil 400 mg PO QD during Part 1 have the option to continue treatment with Belumosudil 400 mg PO QD and subjects randomized to BSC have the option to cross over to treatment with Belumosudil 400 mg PO QD.
  No subject is permitted > 96 weeks of treatment with belumosudil
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belumosudil-R (Experimental): Subjects receive two 200 mg tablets of belumosudil (400 mg) PO QD for 24 weeks. Subjects may also continue treatment with belumosudil 400 mg PO QD after 24 weeks.
  No subject may receive more than 96 weeks of treatment with belumosudil
  Interventions: Drug: Belumosudil
- BSC-R (Active Comparator): Subjects receive best supportive care as determined by the physician. Subjects may later crossover to treatment with belumosudil 400 mg PO QD. No subject may receive more than 96 weeks of treatment with belumosudil.
  Interventions: Other: BSC

INTERVENTIONS:
Drug: Belumosudil
  Other Names: KD025; SLx-2119
  Arms: Belumosudil-R
Other: BSC — Treatment/drug as determined by each subject's prescribing physician
  Other Names: Best standard of care
  Arms: BSC-R

SUMMARY:
This Phase 2 study is to be conducted to evaluate the safety, tolerability, and activity of 400 mg of belumosudil orally (PO) once-daily (QD) compared to Best Supportive Care (BSC) in male and postmenopausal/surgically sterilized female subjects with Idiopathic Pulmonary Fibrosis (IPF). The primary objectives are to evaluate the:

* Change in Forced Vital Capacity (FVC) from baseline to 24 weeks after dosing with belumosudil 400 mg PO QD in subjects with IPF compared to BSC
* Safety and tolerability of belumosudil 400 mg PO QD when administered for 24 weeks to subjects with IPF compared to BSC

DETAILED DESCRIPTION:
Study KD025-207 is a Phase 2, randomized, 2-part, open-label, crossover study in subjects with IPF.

The purpose of the study is to evaluate the safety, tolerability, and activity of 400 mg of belumosudil administered orally (PO) every day (QD) compared to Best Standard of Care (BSC) in subjects with IPF who have previously been treated with or declined treatment with pirfenidone or nintedanib.

The primary objectives are to evaluate the change in Forced Vital Capacity (FVC), and the safety and tolerability from baseline to 24 weeks in subjects with IPF after dosing with belumosudil 400 mg PO QD compared to BSC.

Part 1: Randomized, Open-label for 24 Weeks

Approximately 81 eligible subjects with IPF are to be enrolled, in 10 to 15 sites, and randomized in a 2:1 ratio (belumosudil:BSC) to 1 of the following 2 groups:

* Belumosudil-R (Investigational Group): Belumosudil 400 mg PO QD for 24 weeks
* BSC-R (Control Group): BSC for 24 weeks

The study plan is for 54 subjects to be entered into the Belumosudil-R Treatment Group and 27 subjects into the BSC-R Treatment Group. This sample size provides over 90% power at the 2-sided 0.05 significance level to detect a 20% difference between treatment groups at 24 weeks in percentage change from baseline in FVC assuming a standard deviation (SD) in percentage change from baseline in FVC of 17%. The sample size of 54 subjects receiving belumosudil provides over 90% probability of ≥ 1 subject in the study experiencing an AE that had an underlying rate of ≥ 5%.

Part 2: Continuation of Belumosudil Therapy or Crossover to Belumosudil Therapy Subjects in the Belumosudil-R group who complete 24 weeks of treatment with belumosudil 400 mg PO QD have the option of continuing therapy with belumosudil 400 mg PO QD up to an additional 72 weeks if there are no safety signals and if clinical progress continues. No subject in the Belumosudil-R group is to be permitted to receive therapy with belumosudil greater than a total of 96 weeks.

Subjects in control group BSC-R who complete 24 weeks of BSC have the option of crossing over to therapy with belumosudil 400 mg PO QD for up to 96 weeks if there are no safety signals and if clinical progress continues. No subject in control group BSC-R is to be permitted to receive belumosudil 400 mg PO QD therapy greater than 96 weeks.

Follow-up Period:

Follow-up Visits are to occur 30 days (± 3 days) after the last dose of belumosudil during which subjects are to undergo safety assessments. (A Follow-up Visit is not necessary for subjects receiving BSC.)

Duration of Study for Individual Subjects:

1. Subjects randomized to belumosudil: total up to 104 weeks (4-week screening, 96-week treatment with belumosudil, and 4-week follow-up)
2. Subject randomized to BSC: total up to 128 weeks (4-week screening; up to 24-week treatment with BSC, 96-week treatment with belumosudil, and 4-week follow-up)

Efficacy Assessments

* FVC
* FVC% Predicted
* 6-minute Walking Distance (6MWD)
* Diffusing Capacity of Carbon Monoxide (DLCO)
* Lung Fibrosis (by HRCT and Radiologist's Visual Assessments)
* Time to Acute Exacerbation
* Time to Progression of IPF
* Time to Respiratory-related Hospitalization
* Time to Respiratory-related Death
* St. Georges Respiratory Questionnaire (SGRQ)

Biomarker Assessments

* Matrix Metalloproteinase-7 (MMP7)
* Chemokine Ligand 18 (CCL18)
* Surfactant Protein-D (SPD)

Safety Assessments

* Adverse event (AE)
* Serious adverse event (SAE)
* Physical examination (PE)
* Vital signs (VS)
* Clinical laboratory evaluations (hematology, chemistry, and urinalysis)
* Electrocardiogram (ECG)
* Reason for treatment discontinuation due to toxicity

Analyses

Efficacy and safety are to be analyzed at the end of Part 1 (Week 24) and for the Entire Treatment Period (Parts 1 and 2). Analyses of study subjects are to be grouped and defined as follows:

* Belumosudil-R: subjects randomized to belumosudil
* BSC-R: subjects randomized to BSC
* Belumosudil-WC: subjects randomized to belumosudil plus subjects randomized to BSC and who cross over to treatment with belumosudil
* BSC-NC: subjects randomized to BSC and who cross over to treatment with belumosudil but have data censored by the date of crossover

ELIGIBILITY:
Inclusion Criteria:

A subject had to meet all of the following criteria to be eligible for the study:

1. Adult male and postmenopausal/surgically sterilized female subjects at least 18 years of age (if female, was surgically sterilized [i.e., total hysterectomy, or bilateral salpingo-oophorectomy]).
2. Able to provide written informed consent before the performance of any study specific procedures.
3. IPF diagnosis within 5 years before study entry, proven according to the American Thoracic Society/European Respiratory Society consensus conference criteria, with surgical lung biopsy. In the absence of a surgical lung biopsy, high-resolution computerized tomography (HRCT) consistent with usual interstitial pneumonitis.
4. Resting state pulse oximeter oxygen saturation (SpO2) ≥ 88% with or without supplemental oxygen, Forced Vital Capacity % (FVC%) ≥ 50% normal predicted value, and diffusing capcity (in the lung) of carbon monoxide (DLCO) ≥ 30% normal predicted value at baseline.
5. Men with partners of childbearing potential willing to use 2 medically acceptable methods of contraception during the trial and for 3 months after the last dose of study drug. Effective birth control includes:

   1. Intrauterine device plus 1 barrier method
   2. Stable doses of hormonal contraception for ≥ 3 months (e.g., oral, injectible, implant, transdermal) plus 1 barrier method
   3. 2 barrier methods. Effective barrier methods were male or female condoms, diaphragms, and spermicides (creams or gels containing a chemical to kill sperm)
   4. Vasectomy.
6. Have adequate bone marrow function:

   1. Absolute neutrophil count > 1500/mm^3
   2. Hemoglobin (Hb) > 9.0 g/L
   3. Platelets > 100,000/mm^3
7. Willing to complete all study measurements and assessments in compliance with protocol
8. Had either received pirfenidone and/or nintedanib or offered both treatments (with last dose administered at least 1 month before the expected start of study drug dosing). If either or both pirfenidone and nintedanib treatment had not been given, then documentation that the subject was offered both treatments must have been documented.

Exclusion Criteria:

A subject who met any of the following criteria was ineligible for the study:

1. Interstitial lung disease caused by conditions other than IPF
2. Severe concomitant illness limiting life expectancy (< 1 year)
3. DLCO < 30% predicted
4. Residual volume (RV) ≥ 120% predicted
5. Obstructive lung disease: Forced Expiratory Volume in 1 Second (FEV1/FVC ratio < 0.70)
6. Documented sustained improvement of the subject's IPF condition up to 12 months before study entry with or without IPF-specific therapy
7. Pulmonary infection or upper respiratory tract infection (URTI) within 4 weeks before study entry
8. Acute or chronic impairment (other than dyspnea) limiting the ability to comply with study requirements (e.g., pulmonary function tests [PFTs])
9. Chronic heart failure with New York Heart Association Class III/IV or known left ventricular ejection fraction < 25%
10. Moderate to severe hepatic impairment (i.e., Child-Pugh Class B or C)
11. Estimated creatinine clearance < 30 mL/min
12. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2.0 * upper limit of normal (ULN)
13. Hb < 75% of the lower limit of normal
14. Systolic blood pressure < 100 mmHg
15. Pregnant or breastfeeding female subject
16. Men whose partner is pregnant or breastfeeding
17. Current drug or alcohol dependence
18. Chronic treatment with the following drugs within 4 weeks of study entry and during the study:

    1. Immunosuppressive or cytotoxic drugs including cyclophosphamide and azathioprine
    2. Antifibrotic drugs including pirfenidone, nintedanib, D-penicillamine, colchicine, tumor necrosis factor-alpha blockers, imatinib, and interferon-γ
    3. Chronic use of N-acetylcysteine prescribed for IPF (> 600 mg/day)
    4. Oral anticoagulants prescribed for IPF
19. Treatment with endothelin receptor antagonists within 4 weeks before study entry
20. Systemic treatment within 4 weeks before study entry with cyclosporine A or tacrolimus, everolimus, or sirolimus (calcineurin or mammalian target of rapamycin inhibitors)
21. Previous exposure to belumosudil or known allergy/sensitivity to belumosudil or any other Rho-associated protein kinase 2 (ROCK2) inhibitor
22. Planned treatment or treatment with another investigational drug within 4 weeks before study entry
23. Taking a medication with the potential for QTc prolongation
24. Taking a drug sensitive substrate of CYP enzymes
25. Taking a strong inducer of CYP3A4
26. Had consumed an herbal medication (e.g., St. John's Wort) or grapefruit/grapefruit juice within 14 days prior to the Week 1 Day 1 visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - UC Davis Medical Center, Division of Pulmonary/CC/SM, Sacramento, California
  - St. Francis Medical Institute, Clearwater, Florida
  - Pulmonary Disease Specialists, PA, d/b/a PDS Research, Kissimmee, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Piedmont Healthcare Pulmonary and Critical Care Research, Austell, Georgia
  - Pulmonix, LLC, Greensboro, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 76 unique subjects were randomized in this study. Subjects were randomized to belumosudil 400 mg PO QD or Best Standard of Care (BSC) for first 24 weeks. Subjects were randomized to belumosudil had the option of continuing treatment with belumosudil. No subject in either randomized group were permitted > 96 weeks of treatment. After 24 weeks, subjects randomized to BSC were permitted to crossover to belumosudil; 17 subjects crossed over.
Groups:
- Belumosudil-R: Subjects randomized to treatment with belumosudil 400 mg orally (PO) once daily 9QD).
- BSC-R: Subjects randomized to treatment with best supportive care (BSC) for 24 weeks.
Period: Initial Treatment Period (24 Weeks)
Arm/Group | Belumosudil-R | BSC-R
Started | 52 | 24
Treated | 51 (1 subject was randomized but did not receive treatment.) | 24
Completed | 51 | 18
Not Completed | 1 | 6
Not completed — Death | 0 | 1
Not completed — Cross-overed before Initial Treatment Period (24 Weeks) | 0 | 5
Not completed — Subject was randomized but did not receive treatment | 1 | 0
Period: Post Switch Treatment Period (72 Weeks)
Arm/Group | Belumosudil-R | BSC-R
Started | 51 (51 subjects originally randomized to treatment with belumosudil 400 mg PO QD continued receiving belumosudil 400 mg PO QD.) | 17 (17 subjects randomized to treatment with BSC-R cross-overed to treatment with belumosudil 400 mg PO QD.)
Completed | 23 | 3
Not Completed | 28 | 14
Not completed — Death | 7 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 10 | 6
Not completed — Withdrawal by Subject | 10 | 6

BASELINE CHARACTERISTICS:
Population: One subject randomized to belumosudil 400 mg PO QD did not receive study medication.
  Analysis was performed using the safety population that consisted of all subjects who were randomized and received ≥ 1 dose of belumosudil-R or, for subjects who had BSC, week 1 assessments. Available data at baseline have been reported.
Groups:
- Belumosudil 400 mg PO QD: Randomized to treatment with belumosudil 400 mg (two 200-mg tablets) orally once daily.
- BSC-R: Subjects randomized to treatment with best supportive care for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Belumosudil 400 mg PO QD | BSC-R | Total
Number analyzed (Participants) | 51 | 24 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (7.0) | 74.9 (5.9) | 73.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 38 | 18 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 45 | 24 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 49 | 24 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Prior Use of Pirfenidone [Count of Participants; unit: Participants]
  Yes | 13 | 4 | 17
  No | 38 | 20 | 58
Prior Use of Nintedanib [Count of Participants; unit: Participants]
  Yes | 10 | 4 | 14
  No | 41 | 20 | 61
Prior Use of Pirfenidone or Nintedanib [Count of Participants; unit: Participants]
  Yes | 19 | 6 | 25
  No | 32 | 18 | 50
GAP Stage [Count of Participants; unit: Participants] — GAP = Gender/Age/Physiology. Stage based on total points.
  G: Gender Points: female = 0 points; male = 1 points
  A: Age Points: ≤ 60 years = 0 points; 61-65 years = 1 point; > 65 years = 2 points
  P: Physiology-- FVC% Predicted: > 75% = 0 points; 50-75% = 1 point; ≤ 50% = 2 points DLCO% Predicted: > 55% = 0 points; 36-55% = 1 point; ≤ 35% = 2 points; cannot perform = 3 points
  STAGE
  Stage I Index: 0 to 3 points
  Stage II Index: 4 to 5 points
  Stage III Index: 6 to 8 points
  Participants
    Stage I | 11 | 7 | 18
    Stage II | 31 | 12 | 43
    Stage III | 9 | 5 | 14
Presence of Aggravated Dyspnea Within 6 Months Prior to Informed Consent [Count of Participants; unit: Participants]
  Yes | 18 | 11 | 29
  No | 33 | 13 | 46
Presence of Chest Interstitial Lung Abnormalities Within 6 Months Prior to Informed Consent [Count of Participants; unit: Participants]
  Yes | 23 | 11 | 34
  No | 28 | 13 | 41
SpO2 < 88% Within 6 Months Prior to Informed Consent [Count of Participants; unit: Participants]
  Yes | 7 | 4 | 11
  No | 44 | 20 | 64

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Mean Changes in FVC From Baseline to Week 24
Description: Changes in the mean Forced Vital Capacity (FVC) from baseline at Week 24. Normal FVC-- Healthy males 20 to 60 years: 4.75 to 5.5 L; healthy females 20 to 60 years: 3.25 to 3.75 L
Time Frame: 24 weeks
Population: Analysis was performed using randomized population. Available data for change from baseline at Week 24 have been reported.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Belumosudil-WC: Subjects randomized to treatment with belumosudil 400 mg PO QD plus subjects randomized to treatment with BSC but cross over to treatment with belumosudil 400 mg PO QD
- BSC-NC: Subjects randomized to treatment with BSC and who cross over to treatment with belumosudil 400 mg PO QD but have data censored by the date of crossover
- Total: Subjects randomized to belumosudil 400 mg PO QD plus those randomized to BSC
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 52 | 24 | 69 | 24 | 76
mL
  Baseline: number analyzed (Participants) | 52 | 24 | 64 | 24 | 76
  Baseline | 2608.2 (829.6) | 2516.7 (741.8) | 2608.8 (840.4) | 2516.7 (741.8) | 2569.3 (794.3)
  At Week 24: number analyzed (Participants) | 38 | 21 | 46 | 19 | 59
  At Week 24 | 2626.8 (886.9) | 2438.1 (757.1) | 2617.4 (890.8) | 2436.8 (784.5) | 2533.7 (832.7)
  Change at Week 24: number analyzed (Participants) | 38 | 21 | 46 | 19 | 59
  Change at Week 24 | -115.8 (330.3) | -71.2 (254.2) | -110.8 (316.4) | -103.4 (225.0) | -99.5 (281.4)

2. Primary Outcome: Efficacy: Mean Changes in FVC% Predicted From Baseline at Week 24
Description: Changes in the mean Forced Vital Capacity (FVC)% Predicted from baseline at Week 24.
  Normal FVC%: 80% to 120%
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of predicted
Groups:
- Belumosudil-R: Subjects randomized to treatment with belumosudil 400 mg orally once daily.
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 52 | 24 | 69 | 24 | 76
% of predicted
  Baseline: number analyzed (Participants) | 52 | 24 | 64 | 24 | 76
  Baseline | 69.61 (18.07) | 68.46 (15.63) | 69.73 (17.70) | 68.46 (15.63) | 69.19 (16.71)
  At Week 24: number analyzed (Participants) | 38 | 21 | 46 | 19 | 59
  At Week 24 | 69.71 (19.20) | 68.29 (13.41) | 69.96 (18.43) | 68.58 (13.98) | 69.24 (16.25)
  Change at Week 24: number analyzed (Participants) | 38 | 21 | 46 | 19 | 59
  Change at Week 24 | -2.82 (7.57) | -2.00 (7.36) | -2.66 (7.49) | -3.00 (6.41) | -2.58 (7.16)

3. Primary Outcome: Safety: Percentages of Subjects With Non-serious TEAEs and Relationship to Study Treatment
Description: Percentage of subjects with non-serious TEAEs by relationship to treatment with belumosudil, BSC, or belumosudil and BSC.
  Severity of TEAEs were measured using the Common Terminology Criteria for Adverse Events (CTCAE) version 22.1 (Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = fatal).
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96) of treatment with belumosudil. Subjects randomized to BSC had the option of crossing over at 24 weeks.
Population: All subjects treated in study.
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 51 | 24 | 68 | 24 | 75
Participants
  TEAEs Related to Treatment (All Grades) | 23 | 9 | 32 | 2 | 32
  TEAEs Related to Treatment (Only Grades 3 & 4) | 2 | 0 | 2 | 0 | 2

4. Primary Outcome: Safety: Percentages of Subjects With SAEs Related to Study Treatment
Description: Percentage of subjects with serious TEAEs by relationship to treatment with belumosudil and/or BSC.
  Investigators assessed whether events were related to treatment as possibly, probably, or definitely related.
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96) of treatment with belumosudil. Subjects randomized to BSC and crossing over also up to 24 weeks of BSC.
Population: All subjects treated in study.
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 51 | 24 | 68 | 24 | 75
Participants | 2 | 0 | 2 | 0 | 2

5. Primary Outcome: Safety: Percentages of Subjects With TEAEs Leading to Discontinuation of Treatment With Belumosudil
Description: Percentage of subjects with treatment-emergent adverse events (TEAEs) leading to subjects discontinuing from treatment.
  Investigators assessed whether TEAEs leading to discontinuation were related to study drug (possibly, probably, or definitely), belumosudil 400 mg PO QD.
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96) of treatment with belumosudil
Population: Subjects who received belumosudil 400 mg PO QD were included. Subjects who only received BSC and did not cross over to treatment with belumosudil were not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | Total
Number analyzed (Participants) | 51 | 24 | 68 | 75
Participants
  All TEAEs Leading to Discontinuation | 14 | 8 | 22 | 22
  TEAEs Related to Belumosudil Leading to Study Discontinuation | 5 | 1 | 6 | 6

6. Primary Outcome: Safety: Percentages of Subjects With Deaths Related to Study Treatment
Description: Percentage of subjects with deaths by relationship to treatment with belumosudil, BSC, or belumosudil and BSC.
  Investigators assessed whether events were related to treatment as possibly, probably, or definitely related.
Time Frame: Up to 96 weeks (Weeks 24, 8, and 96) of treatment with belumosudil. Subjects randomized to BSC also had the option of crossing over to treatment with belumosudil at 24 weeks.
Population: All subjects treated in study.
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 51 | 24 | 68 | 19 | 75
Participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Efficacy: Mean Changes in FVC From Baseline at Week 24 by GAP Stage and by Use of Pirfenidone or Nintedanib--
Description: Changes in the mean Forced Vital Capacities (FVC) at Week 24 by Gender/Age/Physiology (GAP) Stage and by the previous use of pirfenidone and/or nintedanib prior to the study for Belumosudil-WC compared to BSC-NC.
  Normal FVC--Healthy males 20 to 60 years: 4.75 to 5.5 L; healthy famles 20 to 60 years: 3.25 to 3.75 L
  GAP is measured by points as follows:
  (G) Gender: Female = 0 points; Male = 1 point (A) Age: ≤ 60 years = 0 points; 61-65 years = 1 point; > 65 years = 2 points (P) Physiology:
  * FVC% Predicted: > 75% = 0 points; 50-75% = 1 point; ≤ 50% = 2 points
  * DLCO% (diffusing lung capacity of carbon monoxide by % predicted) Predicted: > 55% = 0 points; 36-55% = 1 point, ≤ 35% = 2 points; cannot perform = 3 points
  GAP Stage:
  * Stage I Index = 0 to 3 points
  * Stage II Index= 4 to 5 points
  * Stage III Index = 6 to 8 points
Time Frame: 24 weeks
Population: The Modified Intent-to-Treat (mITT) Population was used which consisted of all subjects in the Safety Population who had an evaluable baseline and ≥ 1 evaluable post baseline assessment.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Belumosudil-WC | BSC-NC
Number analyzed (Participants) | 58 | 21
mL
  GAP Stage I: number analyzed (Participants) | 13 | 7
  GAP Stage I | -117.65 [-324.28 to 88.98] | -156.50 [-355.39 to 42.40]
  GAP Stage II: number analyzed (Participants) | 26 | 9
  GAP Stage II | -219.90 [-416.20 to -23.60] | -179.94 [-444.35 to 84.47]
  GAP Stage III: number analyzed (Participants) | 7 | 3
  GAP Stage III | 101.95 [-1246.61 to 1450.50] | 7.79 [-1553.37 to 1568.95]
  No Prior Use of Pirfenidone or Nintedanib: number analyzed (Participants) | 34 | 16
  No Prior Use of Pirfenidone or Nintedanib | -80.34 [-190.81 to 30.14] | -46.21 [-167.93 to 75.51]
Statistical Analysis 1: Comparison: Belumosudil-WC vs BSC-NC; GAP Stage I-- Difference: Belumosudil-WC minus BSC-NC = 38.85 (95% CI: -126.99, 204.69) mL; Test type: Superiority; p = 0.5733, Mixed Models Analysis; Results are not stable due to small sample size and signal/noise ratio
Statistical Analysis 2: Comparison: Belumosudil-WC vs BSC-NC; GAP Stage II-- Difference: Belumosudil-WC minus BSC-NC = -39.96 (95% CI: -288.63, 208.71) mL; Test type: Superiority; p = 0.6967, Mixed Models Analysis; Results are not stable due to small sample size and signal/noise ratio
Statistical Analysis 3: Comparison: Belumosudil-WC vs BSC-NC; GAP Stage III-- Difference: Belumosudil-WC minus BSC-NC = 94.16 (95% CI: -1103.56, 1291.88) mL; Test type: Superiority; p = 0.5003, Mixed Models Analysis; Results are not stable due to small sample size and signal/noise ratio
Statistical Analysis 4: Comparison: Belumosudil-WC vs BSC-NC; No Prior Pirfenidone or Nintedanib-- Difference: Belumosudil-WC minus BSC-NC = -34.13 (95% CI: -137.08, 68.82); Test type: Superiority; p = 0.4866, Mixed Models Analysis; Results are not stable due to small sample size and signal/noise ratio

8. Secondary Outcome: Efficacy: Mean Changes in FVC From Baseline at Week 48, Week 96, and EOT
Description: Changes in the mean Forced Vital Capacity (FVC) from baseline at Weeks 48 and 96, and End-of-Treatment (EOT) Normal FVC: Healthy males 20 to 60 years: 4.75 to 5.25 L; healthy females 20 to 60 years: 3.25 to 3.75 L
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | Total
Number analyzed (Participants) | 52 | 24 | 69 | 76
mL
  Baseline: number analyzed (Participants) | 52 | 24 | 64 | 76
  Baseline | 2608.2 (829.6) | 2516.7 (741.8) | 2608.8 (840.4) | 2569.3 (794.3)
  Change at Week 48: number analyzed (Participants) | 29 | 8 | 35 | 37
  Change at Week 48 | -197.2 (331.5) | -82.5 (329.7) | -199.6 (366.1) | -177.8 (358.8)
  Change at Week 96: number analyzed (Participants) | 20 | 5 | 23 | 25
  Change at Week 96 | -141.0 (401.1) | -264.0 (896.0) | -122.2 (384.3) | -147.5 (492.3)
  Change at EOT: number analyzed (Participants) | 21 | 7 | 27 | 28
  Change at EOT | -227.9 (367.7) | -110.7 (397.7) | -207.2 (353.7) | -180.9 (355.8)

9. Secondary Outcome: Efficacy: Mean Change in Mean FEV1/FVC Ratio From Baseline at Weeks 24, 48, and 96 and EOT
Description: Change in the mean ratio of Forced Expiratory Volume in 1 Second (FEV1) divided by the Forced Vital Capacity (FVC) at Week 24, Week 48, Week 96, and End-of-Treatment (EOT) Normal FEV1: 80% to 120% FEV1/FVC = Within 5% of predicted ratio
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 52 | 24 | 69 | 24 | 76
Units
  Baseline: number analyzed (Participants) | 52 | 24 | 64 | 24 | 76
  Baseline | 0.829 (0.0613) | 0.816 (0.0674) | 0.832 (0.0584) | 0.816 (0.0674) | 0.825 (0.0623)
  Change at Week 24: number analyzed (Participants) | 38 | 21 | 46 | 19 | 59
  Change at Week 24 | -0.006 (0.0444) | 0.013 (0.0310) | -0.005 (0.0410) | 0.016 (0.0311) | 0.004 (0.0378)
  Change at Week 48: number analyzed (Participants) | 29 | 8 | 35 | 0 | 37
  Change at Week 48 | 0.001 (0.0251) | -0.005 (0.0141) | -0.001 (0.0249) |  | -0.002 (0.0232)
  Change at Week 96: number analyzed (Participants) | 20 | 5 | 23 | 0 | 25
  Change at Week 96 | -0.012 (0.0420) | -0.014 (0.0378) | -0.012 (0.0402) |  | -0.012 (0.0391)
  Change at EOT: number analyzed (Participants) | 21 | 7 | 27 | 1 | 28
  Change at EOT | -0.010 (0.0362) | 0.011 (0.0372) | -0.011 (0.0453) | -0.010 (0) | -0.007 (0.0436)

10. Secondary Outcome: Efficacy: Mean Changes in FVC% Predicted at Week 24 by GAP Stage and by Use of Pirfenidone or Nintedanib--
Description: Changes in the mean Forced Vital Capacities (FVC)% Predicted at Week 24 by Gender/Age/Physiology (GAP) Stage and by the previous use of pirfenidone and/or nintedanib prior to the study for Belumosudil-WC compared to BSC-NC.
  GAP is measured by points as follows:
  (G) Gender: Female = 0 points; Male = 1 point (A) Age: ≤ 60 years = 0 points; 61-65 years = 1 point; > 65 years = 2 points (P) Physiology:
  * FVC% Predicted: > 75% = 0 points; 50-75% = 1 point; ≤ 50% = 2 points
  * DLCO% (diffusing lung capacity of carbon monoxide by % predicted) Predicted: > 55% = 0 points; 36-55% = 1 point, ≤ 35% = 2 points; cannot perform = 3 points
  GAP Stage:
  * Stage I = 0 to 3 points
  * Stage II = 4 to 5 points
  * Stage III = 6 to 8 points
Time Frame: 24 weeks
Population: as for outcome 7
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: % of predicted
Arm/Group | Belumosudil-WC | BSC-NC
Number analyzed (Participants) | 58 | 21
% of predicted
  GAP Stage I: number analyzed (Participants) | 13 | 7
  GAP Stage I | -4.65 [-11.34 to 2.03] | -6.53 [-13.14 to 0.07]
  GAP Stage II: number analyzed (Participants) | 26 | 9
  GAP Stage II | -6.42 [-11.69 to -1.15] | -4.69 [-11.58 to 2.19]
  GAP Stage III: number analyzed (Participants) | 7 | 3
  GAP Stage III | 2.34 [-36.32 to 40.99] | -0.15 [-42.95 to 42.65]
  Prior Use of Pirfenidone or Nintedanib: number analyzed (Participants) | 12 | 3
  Prior Use of Pirfenidone or Nintedanib | -6.20 [-58.23 to 45.82] | -14.91 [-92.49 to 62.68]
Statistical Analysis 1: Comparison: Belumosudil-WC vs BSC-NC; Test type: Superiority — GAP Stage I-- Difference: Belumosudil-WC minus BSC-NC = 1.88 (95% CI: -2.69, 6.45); p = 0.3391, Mixed Models Analysis; Results are not stable due to small sample size and signal/noise ratio
Statistical Analysis 2: Comparison: Belumosudil-WC vs BSC-NC; Test type: Superiority — GAP Stage II-- Difference: Belumosudil-WC minus BSC-NC = -1.72 (95% CI: -8.13, 4.69); p = 0.5201, Mixed Models Analysis; Results are not stable due to small sample size and signal/noise ratio
Statistical Analysis 3: Comparison: Belumosudil-WC vs BSC-NC; Test type: Superiority — GAP Stage III-- Difference: Belumosudil-WC minus BSC-NC = 2.48 (95% CI: -23.84, 28.81); p = 0.4426, Mixed Models Analysis; Results are not stable due to small sample size and signal/noise ratio
Statistical Analysis 4: Comparison: Belumosudil-WC vs BSC-NC; Test type: Superiority — No Prior Use of Pirfenidone or Nintedanib-- Difference: Belumosudil-WC minus BSC-NC = 8.70 (95% CI: -78.76, -96.17); p = 0.4260, Mixed Models Analysis; Results are not stable due to small sample size and signal/noise ratio

11. Secondary Outcome: Efficacy: Percentages of Subjects With Decrease ≥ 5% in FVC% Predicted From Baseline at Weeks 24, 48, and 96
Description: Percentage of subjects exhibiting at least a 5% decrease in Forced Vital Capacity (FVC)% Predicted from baseline at Week 24, at Week 48, and at Week 96
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 46 | 24 | 58 | 21 | 70
Participants
  At Week 24: Yes: number analyzed (Participants) | 38 | 21 | 46 | 19 | 59
  At Week 24: Yes | 11 | 7 | 14 | 7 | 21
  At Week 24: No: number analyzed (Participants) | 38 | 21 | 46 | 19 | 59
  At Week 24: No | 27 | 14 | 32 | 12 | 42
  At Week 48: Yes: number analyzed (Participants) | 29 | 8 | 35 | 0 | 37
  At Week 48: Yes | 14 | 4 | 16 |  | 18
  At Week 48: No: number analyzed (Participants) | 29 | 8 | 35 | 0 | 37
  At Week 48: No | 15 | 4 | 19 |  | 20
  At Week 96: Yes: number analyzed (Participants) | 20 | 5 | 23 | 0 | 25
  At Week 96: Yes | 6 | 2 | 6 |  | 8
  At Week 96: No: number analyzed (Participants) | 20 | 5 | 23 | 0 | 25
  At Week 96: No | 14 | 3 | 17 |  | 17

12. Secondary Outcome: Efficacy: Percentage of Subjects With Decrease ≥ 10% in FVC% Predicted at Weeks 24, 48, and 96
Description: Percentage of subjects who exhibited at least a 10% decrease in Forced Vital Capacity (FVC)% Predicted from baseline at Week 24, at Week 48, and at Week 96
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 46 | 24 | 58 | 21 | 70
Participants
  At Week 24: Yes: number analyzed (Participants) | 38 | 21 | 46 | 19 | 59
  At Week 24: Yes | 5 | 4 | 6 | 4 | 10
  At Week 24: No: number analyzed (Participants) | 38 | 21 | 46 | 19 | 59
  At Week 24: No | 33 | 17 | 40 | 15 | 50
  At Week 48: Yes: number analyzed (Participants) | 29 | 8 | 35 | 0 | 37
  At Week 48: Yes | 7 | 1 | 9 |  | 10
  At Week 48: No: number analyzed (Participants) | 29 | 8 | 35 | 0 | 37
  At Week 48: No | 22 | 7 | 26 |  | 30
  At Week 96: Yes: number analyzed (Participants) | 20 | 5 | 23 | 0 | 25
  At Week 96: Yes | 5 | 2 | 5 |  | 7
  At Week 96: No: number analyzed (Participants) | 20 | 5 | 23 | 0 | 25
  At Week 96: No | 15 | 3 | 18 |  | 18

13. Secondary Outcome: Efficacy: Mean Change in 6MWD at Weeks 24, 48, and 96
Description: The mean change in the 6-mile Walking Distance (6MWD), i.e., the distance a subject can walk in 6 minutes, from baseline to Week 24, to Week 48, and to Week 96.
  Positive change = improvement; negative change = worsening
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 52 | 24 | 69 | 24 | 76
meters
  Baseline: number analyzed (Participants) | 51 | 24 | 65 | 19 | 75
  Baseline | 368.59 (168.84) | 349.25 (180.40) | 350.12 (168.88) | 323.11 (126.64) | 345.17 (163.88)
  Change at Week 24: number analyzed (Participants) | 37 | 20 | 45 | 13 | 57
  Change at Week 24 | -12.11 (101.78) | -16.60 (66.80) | 7.53 (177.88) | -0.77 (49.08) | -0.04 (140.22)
  Change at Week 48: number analyzed (Participants) | 30 | 8 | 36 | 0 | 38
  Change at Week 48 | -18.33 (102.45) | 119.00 (364.61) | -18.83 (95.33) |  | 6.23 (178.69)
  Change at Week 96: number analyzed (Participants) | 17 | 5 | 20 | 0 | 22
  Change at Week 96 | -23.06 (78.84) | -47.80 (69.80) | -20.98 (72.80) |  | -26.34 (71.60)

14. Secondary Outcome: Efficacy: Percentages of Subjects With ≥ 50 Meter Improvement in 6MWD at Weeks 24, 48, and 96
Description: The percentage of subjects who have at least a 50 meter improvement in the 6-mile Walking Distance (6MWD), i.e., the distance a subject can walk in 6 minutes, from baseline to Week 24, Week 48, and Week 96.
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 46 | 24 | 58 | 21 | 70
Participants
  ≥ 50 Meter Improvement at Week 24: Yes: number analyzed (Participants) | 37 | 20 | 45 | 13 | 57
  ≥ 50 Meter Improvement at Week 24: Yes | 6 | 4 | 8 | 2 | 11
  ≥ 50 Meter Improvement at Week 24: No: number analyzed (Participants) | 37 | 20 | 45 | 13 | 70
  ≥ 50 Meter Improvement at Week 24: No | 31 | 16 | 37 | 11 | 48
  ≥ 50 Meter Improvement at Week 48: Yes: number analyzed (Participants) | 30 | 8 | 36 | 0 | 38
  ≥ 50 Meter Improvement at Week 48: Yes | 6 | 2 | 8 |  | 10
  ≥ 50 Meter Improvement at Week 48: No: number analyzed (Participants) | 30 | 8 | 36 | 0 | 38
  ≥ 50 Meter Improvement at Week 48: No | 24 | 6 | 28 |  | 32
  ≥ 50 Meter Improvement at Week 96: Yes: number analyzed (Participants) | 17 | 5 | 20 | 0 | 22
  ≥ 50 Meter Improvement at Week 96: Yes | 5 | 2 | 5 |  | 7
  ≥ 50 Meter Improvement at Week 96: No: number analyzed (Participants) | 17 | 5 | 20 | 0 | 22
  ≥ 50 Meter Improvement at Week 96: No | 12 | 3 | 15 |  | 15

15. Secondary Outcome: Efficacy: Mean Changes in DLCO (%) at Weeks 24, 48, and 96
Description: The diffusing capacity for carbon dioxide (DLCO) is a measure of the conductance of gas transfer from inspired gas to the red blood cells.
  Normal DLCO is > 75% of predicted up to 140%. Severity is generally rated as:
  * Mild: 60% to lower limit of normal
  * Moderate: 40% to 60%
  * Severe: < 40%
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: % of diffusing capacity of CO
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 52 | 24 | 69 | 24 | 76
% of diffusing capacity of CO
  Baseline: number analyzed (Participants) | 51 | 24 | 63 | 19 | 75
  Baseline | 47.3 (11.7) | 47.3 (9.9) | 47.1 (12.0) | 48.0 (10.2) | 47.3 (11.1)
  Change at Week 24: number analyzed (Participants) | 35 | 21 | 42 | 15 | 56
  Change at Week 24 | -2.7 (9.5) | -3.8 (5.4) | -3.1 (9.3) | -4.5 (5.6) | -3.6 (7.7)
  Change at Week 48: number analyzed (Participants) | 28 | 8 | 34 | 0 | 36
  Change at Week 48 | -2.9 (8.3) | -7.1 (12.7) | -3.2 (8.0) |  | -3.9 (9.0)
  Change at Week 96: number analyzed (Participants) | 10 | 5 | 13 | 0 | 15
  Change at Week 96 | -4.2 (11.3) | -13.7 (17.7) | -6.0 (11.4) |  | -8.2 (13.4)

16. Secondary Outcome: Efficacy: Percentages of Subjects With Change From Baseline in DLCO (%) ≤ -15% at Weeks 24, 48, and 96
Description: Percentage of the number of subjects who exhibit less than a -15% decrease in diffusing capacity of carbon monoxide (DLCO), measured as % from baseline at Week 24, Week 48, and Week 96
  The diffusing capacity for carbon dioxide (DLCO) is a measure of the conductance of gas transfer from inspired gas to the red blood cells.
  Normal DLCO is > 75% of predicted up to 140%. Severity is generally rated as:
  * Mild: 60% to lower limit of normal
  * Moderate: 40% to 60%
  * Severe: < 40%
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 46 | 24 | 58 | 21 | 70
Participants
  Week 24 Change ≤ -15%: Yes: number analyzed (Participants) | 36 | 21 | 43 | 15 | 57
  Week 24 Change ≤ -15%: Yes | 7 | 7 | 10 | 6 | 16
  Week 24 Change ≤ -15%: No: number analyzed (Participants) | 36 | 21 | 43 | 15 | 57
  Week 24 Change ≤ -15%: No | 29 | 14 | 33 | 9 | 43
  Week 48 Change ≤ -15%: Yes: number analyzed (Participants) | 28 | 8 | 34 | 0 | 36
  Week 48 Change ≤ -15%: Yes | 10 | 4 | 11 |  | 14
  Week 48 Change ≤ -15%: No: number analyzed (Participants) | 28 | 8 | 34 | 0 | 36
  Week 48 Change ≤ -15%: No | 18 | 4 | 23 |  | 24
  Week 96 Change ≤ -15%: Yes: number analyzed (Participants) | 10 | 5 | 13 | 0 | 15
  Week 96 Change ≤ -15%: Yes | 3 | 4 | 5 |  | 7
  Week 96 Change ≤ -15%: No: number analyzed (Participants) | 10 | 5 | 13 | 0 | 15
  Week 96 Change ≤ -15%: No | 7 | 1 | 8 |  | 8

17. Secondary Outcome: Efficacy: Mean Changes in Total Lung Fibrosis Score, by HRCT, From Baseline at Weeks 24, 48, and 96
Description: The change in Total Lung Fibrosis mean score from baseline at Weeks 24, 48, and 96. Measurements using quantitative high-resolution computerized tomography (HRCT) and include (1) extent of fibrotic abnormality; (2) fibrosis score; (3) ground glass opacity; (4) honeycombing score; (5) kurtosis of lung voxel intensity; (6) skewness of lung voxel intensity; (7) standard deviation of voxel; (8) CT total lung volume; (9) normal lung; (10) reticular score; and (11) evaluation of change on sequential scans.
  The Quantitative Lung Fibrosis (QLF) score measures the extent of reticular patterns with architectural distortion due to fibrosis using a support vector machine classifier. Range: 0 to 100. Higher scores imply greater impairment.
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: The mITT Population was used which consisted of all subjects in the Safety Population who had an evaluable baseline and ≥ 1 evaluable post baseline FVC assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 52 | 24 | 69 | 24 | 76
score on a scale
  Baseline: number analyzed (Participants) | 43 | 21 | 45 | 21 | 64
  Baseline | 30.91 (14.54) | 33.34 (17.81) | 31.78 (15.48) | 33.34 (17.81) | 32.53 (16.45)
  Change at Week 24: number analyzed (Participants) | 32 | 17 | 34 | 16 | 49
  Change at Week 24 | 7.36 (11.46) | 1.08 (6.31) | 8.00 (12.55) | 1.41 (6.31) | 4.67 (10.44)
  Change at Week 48: number analyzed (Participants) | 22 | 7 | 23 | 0 | 29
  Change at Week 48 | 6.51 (11.76) | 6.23 (13.27) | 6.01 (11.74) |  | 6.06 (11.87)
  Change at Week 96: number analyzed (Participants) | 15 | 3 | 15 | 0 | 18
  Change at Week 96 | 6.36 (10.41) | 8.47 (21.86) | 6.36 (10.41) |  | 6.71 (12.09)

18. Secondary Outcome: Efficacy: Categorical Changes in Lung Fibrosis as Observed by Sequential Scans of Radiologist Visual Assessment, From Baseline at Weeks 24, 48, and 96
Description: The categorical changes of lung fibrosis using subjective visual assessments by radiologists from sequential scans at baseline, Week 24, Week 48, and Week 96. Changes were categorized as: (1) much better; (2) slightly better; (3) same; (4) slightly worse; and (5) much worse. This categorization is simplified as Better (Much or Slightly); Same; and Worse (Slightly or Much).
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: All randomized subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 46 | 24 | 58 | 21 | 70
Participants
  Week 24: Better: number analyzed (Participants) | 35 | 18 | 43 | 16 | 53
  Week 24: Better | 0 | 1 | 1 | 1 | 1
  Week 24: Same: number analyzed (Participants) | 35 | 18 | 43 | 16 | 53
  Week 24: Same | 22 | 13 | 25 | 11 | 35
  Week 24: Worse: number analyzed (Participants) | 35 | 18 | 43 | 16 | 53
  Week 24: Worse | 13 | 4 | 17 | 4 | 17
  Week 48: Better: number analyzed (Participants) | 16 | 7 | 20 | 0 | 23
  Week 48: Better | 0 | 1 | 1 |  | 1
  Week 48: Same: number analyzed (Participants) | 16 | 7 | 20 | 0 | 23
  Week 48: Same | 6 | 1 | 6 |  | 7
  Week 48: Worse: number analyzed (Participants) | 16 | 7 | 20 | 0 | 23
  Week 48: Worse | 10 | 5 | 13 |  | 15
  Week 96: Better: number analyzed (Participants) | 4 | 2 | 5 | 0 | 6
  Week 96: Better | 0 | 1 | 1 | 0 | 1
  Week 96: Same: number analyzed (Participants) | 4 | 2 | 5 | 0 | 6
  Week 96: Same | 1 | 0 | 1 | 0 | 1
  Week 96: Worse: number analyzed (Participants) | 4 | 2 | 5 | 0 | 6
  Week 96: Worse | 3 | 1 | 3 |  | 4

19. Secondary Outcome: Efficacy: Changes in Mean DTA Lung Fibrosis Score, by Radiologist Visual Assessment, From Baseline at Weeks 24, 48, and 96
Description: The change in Data-driven Texture Analysis (DTA) Lung Fibrosis mean score using sequential scans from Radiologist's Visual Reads from baseline to Weeks 24, 48, and 96. The change in DTA Lung Fibrosis mean score was measured using sequential scans from Radiologist's Visual Reads from baseline at Weeks 24, 48, and 96. DTA fibrosis score was computed as the number of Region of Interests (ROIs) classified as fibrotic divided by the total number of ROIs sampled from the lung segmentation volume. The DTA fibrosis score ranged from 0 - 100%, where higher scores indicated worsening of disease.
Time Frame: Up to 96 Weeks (Weeks 24, 48, and 96)
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: units on a scale (0-100)
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 52 | 24 | 69 | 24 | 76
units on a scale (0-100)
  Baseline: number analyzed (Participants) | 42 | 22 | 48 | 22 | 65
  Baseline | 23.1 (11.99) | 22.7 (10.77) | 22.3 (12.07) | 22.7 (10.77) | 22.5 (11.35)
  Change at Week 24: number analyzed (Participants) | 31 | 17 | 34 | 16 | 48
  Change at Week 24 | 0.3 (4.82) | 0.6 (4.29) | 1.2 (6.86) | 0.6 (4.43) | 0.9 (5.70)
  Change at Week 48: number analyzed (Participants) | 13 | 7 | 14 | 0 | 20
  Change at Week 48 | 3.1 (7.51) | 2.9 (4.88) | 2.9 (7.26) |  | 2.9 (6.44)
  Change at Week 96: number analyzed (Participants) | 4 | 2 | 4 | 0 | 6
  Change at Week 96 | 7.5 (9.57) | 5.0 (7.07) | 7.5 (9.57) |  | 6.7 (8.16)

20. Secondary Outcome: Efficacy: Event-free Probability of Acute Exacerbation of IPF
Description: Acute exacerbation of IPF was defined by the following symptoms within 1 month that could not be explained by other reasons: (1) aggravated dyspnea; (2) newly discovered chest interstitial lung abnormality (by radiograph or HRCT); (3) SpO2 decrease to < 88%.
  Acute exacerbation was diagnosed if Items #1 and #2 were present or if Items #1 and #3 were present and the following AEs did not occur: (A) any AE with the Preferred Term containing the word "infection" or "cardiac failure"; (B) pulmonary embolism; (C) pneumothorax.
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Event-free Probability
Arm/Group | Belumosudil-R | Belumosudil-WC | BSC-NC
Number analyzed (Participants) | 46 | 58 | 21
Event-free Probability
  24 weeks | 0.91 [0.78 to 0.97] | 0.91 [0.80 to 0.96] | 0.92 [0.54 to 0.99]
  48 weeks: number analyzed (Participants) | 46 | 58 | 0
  48 weeks | 0.85 [0.70 to 0.93] | 0.84 [0.70 to 0.92] |
  96 weeks: number analyzed (Participants) | 46 | 58 | 0
  96 weeks | 0.64 [0.44 to 0.78] | 0.66 [0.48 to 0.79] |
Statistical Analysis 1: Comparison: Belumosudil-R vs BSC-NC; Hazard ratio: 0.86 (0.16, 4.48); Test type: Superiority — Cox Regression; p = 0.8561, Log Rank
Statistical Analysis 2: Comparison: Belumosudil-WC vs BSC-NC; Hazard ratio: 0.87 (95% CI: 0.17, 4.33); Test type: Superiority — Cox Regression; p = 0.8608, Log Rank

21. Secondary Outcome: Efficacy: Event-free Probability of Progression of IPF
Description: Progression of IPF exacerbation was defined as the probability of a subject exhibiting IPF time from baseline to any of the following: (1) probability of first respiratory-related hospitalization; (2) probability of respiratory-related death; absolute decline in FVC% Predicted value of ≥ 10% vs. FVC %; probability of predicted value recorded at baseline; and (4) probability of absolute decline in DLCO, adjusted for hemoglobin (Hb), Percent of predicted value of ≥ 15% vs. DLCO at baseline. Subjects randomized to and received BSC were censored on crossover.
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Event-free Probability
Arm/Group | Belumosudil-R | Belumosudil-WC | BSC-NC
Number analyzed (Participants) | 46 | 58 | 21
Event-free Probability
  24 weeks | 0.86 [0.71 to 0.93] | 0.80 [0.67 to 0.88] | 0.66 [0.39 to 0.83]
  48 weeks: number analyzed (Participants) | 46 | 58 | 0
  48 weeks | 0.52 [0.35 to 0.66] | 0.47 [0.33 to 0.60] |
  96 weeks: number analyzed (Participants) | 46 | 58 | 0
  96 weeks | 0.20 [0.09 to 0.35] | 0.16 [0.07 to 0.28] |
Statistical Analysis 1: Comparison: Belumosudil-R vs BSC-NC; Hazard ratio: 0.34 (95% CI: 0.14, 0.79); Test type: Superiority — Cox Regression; p = 0.0084, Log Rank
Statistical Analysis 2: Comparison: Belumosudil-WC vs BSC-NC; Hazard Ratio: 0.47 (95% CI: 0.22, 1.03); Test type: Superiority — Cox Regression; p = 0.0508, Log Rank

22. Secondary Outcome: Efficacy: Event-free Probability of First Respiratory-related Hospitalization
Description: Probability of first-related hospitalization defined as any AE where the high-level group term contained the terms "respiratory" and the AE resulted in a hospitalization. Subjects randomized and received BSC were censored on crossover.
  Note: The hazard ratios for Belumosudil-R vs. BSC-NC and for Belumosudil-WC vs. BSC-NC were not calculable.
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: Analysis was of the Modified Intent-to-Treat (mITT) Population, defined as consisting of all subjects in the Safety Population who had an evaluable baseline and ≥ 1 evaluable post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: Event-free Probability
Arm/Group | Belumosudil-R | Belumosudil-WC
Number analyzed (Participants) | 46 | 58
Event-free Probability
  24 weeks | 0.98 [0.85 to 1.00] | 0.96 [0.86 to 0.99]
  48 weeks | 0.89 [0.74 to 0.96] | 0.85 [0.72 to 0.93]
  96 weeks | 0.79 [0.61 to 0.90] | 0.75 [0.58 to 0.85]

23. Secondary Outcome: Efficacy: Event-free Probability of Respiratory-related Death
Description: Probability of respiratory-related death, defined as any AE where the high-level group term contained the term "respiratory" and the AE resulted in a death.
  Subjects randomized to and who received BSC were censored on crossover.
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: Event-free Probability
Arm/Group | Belumosudil-R | Belumosudil-WC | BSC-NC
Number analyzed (Participants) | 46 | 58 | 21
Event-free Probability
  24 weeks | 0.98 [0.85 to 1.00] | 0.98 [0.87 to 1.00] | 0.95 [0.69 to 0.99]
  48 weeks: number analyzed (Participants) | 46 | 58 | 0
  48 weeks | 0.92 [0.76 to 0.97] | 0.91 [0.77 to 0.97] |
  96 weeks: number analyzed (Participants) | 46 | 58 | 0
  96 weeks | 0.88 [0.71 to 0.95] | 0.88 [0.72 to 0.95] |
Statistical Analysis 1: Comparison: Belumosudil-R vs BSC-NC; Hazard ratio: 0.34 (95% CI: 0.02, 5.54); Test type: Superiority — Cox Regression; p = 0.4251, Log Rank
Statistical Analysis 2: Comparison: Belumosudil-WC vs BSC-NC; Hazard ratio: 0.27 (95% CI: 0.02, 4.45); Test type: Superiority — Cox Regression; p = 0.3294, Log Rank

24. Secondary Outcome: Efficacy: Mean Changes in SGRQ From Baseline at Weeks 24, 48 and 96
Description: The St. George's Respiratory Questionnaire (SGRQ) is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in subjects with obstructive airways disease consisting of 2 parts: (1) symptoms component (frequency & severity) with a 3-month recall; and (2) activities that cause or are limited by breathlessness. Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall.
  Changes were assessed from baseline at Week 24, at Week 48, and at Week 96.
  The SGRQ scores range from 0 to 100, with higher scores indicating greater limitations. Based on empirical data and interviews with subjects, a mean change score of 4 units is associated with slightly efficacious treatment, 8 units for moderately efficacious change, and 12 units for very efficacious treatment
Time Frame: Up to 96 weeks (Weeks 24, 48, and 96)
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
Number analyzed (Participants) | 52 | 24 | 69 | 24 | 76
units on a scale
  Baseline: number analyzed (Participants) | 27 | 12 | 37 | 12 | 42
  Baseline | 64.45 (18.98) | 74.45 (18.94) | 64.86 (18.29) | 74.45 (18.94) | 68.63 (18.83)
  Change at Week 24: number analyzed (Participants) | 31 | 16 | 39 | 15 | 49
  Change at Week 24 | -5.78 (17.74) | -2.64 (9.59) | -2.63 (18.38) | -2.64 (9.59) | -2.64 (14.79)
  Change at Week 48: number analyzed (Participants) | 17 | 3 | 20 | 0 | 21
  Change at Week 48 | 0.36 (15.34) | 2.07 (9.90) | 0.41 (14.63) |  | 0.63 (13.93)
  Change at Week 96: number analyzed (Participants) | 10 | 2 | 11 | 0 | 13
  Change at Week 96 | 1.50 (16.61) | 9.35 (4.54) | 1.37 (15.76) |  | 2.60 (14.75)

ADVERSE EVENTS:
Time Frame: Subjects randomized to belumosudil 400 mg PO QD: up to 96 weeks of treatment Subjects randomized to BSC: 24 weeks of BSC plus up to 96 weeks of treatment with belumosudil 400 mg PO QD
Arm/Group | Belumosudil-R | BSC-R | Belumosudil-WC | BSC-NC | Total
All-Cause Mortality (participants affected / at risk) | 7/51 | 3/24 | 9/68 | 1/24 | 10/75
Serious Adverse Events (participants affected / at risk) | 29/51 | 10/24 | 38/68 | 4/24 | 39/75
Other Adverse Events (participants affected / at risk) | 50/51 | 23/24 | 67/68 | 19/24 | 73/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belumosudil-R (N=51) | BSC-R (N=24) | Belumosudil-WC (N=68) | BSC-NC (N=24) | Total (N=75)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 8 | 1 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 6 | 0 | 6
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Congestive cardiac failure (Cardiac disorders) | 3 | 0 | 3 | 0 | 3
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Acute myocardial infarction (AMI) (Cardiac disorders) | 1 | 2 | 2 | 1 | 3
Anginal equivalent (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 3 | 0 | 3
Complete atrioventricular block (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1 | 2 | 1 | 2
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Myocardial infarction (MI) (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 0 | 4 | 0 | 4
Corona virus infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Pneumona influenzal (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 1 | 1
Localized infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Viral pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 1
Chills (General disorders) | 1 | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Melena (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 2
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Basal ganglia hemorrhage (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Transient ischemic attack (TIA) (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Troponin increased (Investigations) | 1 | 0 | 1 | 0 | 1
Abnormal urine analysis (Investigations) | 1 | 0 | 1 | 0 | 1
Metastatic lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 2 | 0 | 2
Superficial thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Hypovolemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1
Toe amputation (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 1
Lung transplant (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 1
Amaurosis fugax (Eye disorders) | 0 | 1 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belumosudil-R (N=51) | BSC-R (N=24) | Belumosudil-WC (N=68) | BSC-NC (N=24) | Total (N=75)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 | 5 | 21 | 4 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 14 | 8 | 22
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 8 | 1 | 9
Exertional dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 1 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 2 | 5
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5 | 0 | 5
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0 | 3
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 2
Upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 0 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2
Sputum discolored (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 8 | 5 | 11 | 2 | 13
Bronchitis (Infections and infestations) | 7 | 5 | 7 | 5 | 12
Pneumonia (Infections and infestations) | 7 | 0 | 7 | 0 | 7
Upper respiratory tract infection (Infections and infestations) | 5 | 6 | 8 | 4 | 11
Viral gastroenteritis (Infections and infestations) | 4 | 0 | 4 | 0 | 4
Sinusitis (Infections and infestations) | 3 | 0 | 3 | 0 | 3
Tooth infection (Infections and infestations) | 3 | 0 | 3 | 0 | 3
Cellulitis (Infections and infestations) | 2 | 2 | 4 | 1 | 4
Corona virus infection (Infections and infestations) | 2 | 0 | 2 | 0 | 2
Influenza (Infections and infestations) | 2 | 1 | 3 | 0 | 3
Rhinitis (Infections and infestations) | 2 | 1 | 3 | 0 | 3
Urinary tract infection (Infections and infestations) | 2 | 1 | 2 | 1 | 3
Viral infection (Infections and infestations) | 2 | 0 | 2 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 12 | 6 | 18 | 0 | 18
Nausea (Gastrointestinal disorders) | 6 | 4 | 8 | 3 | 10
Upper abdominal pain (Gastrointestinal disorders) | 3 | 1 | 4 | 0 | 4
Constipation (Gastrointestinal disorders) | 3 | 1 | 4 | 0 | 4
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2
Gastroesophageal reflux disease (GERD) (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 2
Alanine aminotransferase (ALT) increased (Investigations) | 8 | 3 | 10 | 1 | 11
Aspartate aminotransferase (AST) increased (Investigations) | 6 | 2 | 8 | 0 | 8
Gamma-glutamyltransferase (GGT) increased (Investigations) | 5 | 3 | 6 | 2 | 8
Blood creatinine increased (Investigations) | 3 | 1 | 3 | 1 | 4
Prothrombin time prolonged (Investigations) | 2 | 0 | 2 | 0 | 2
Weight decreased (Investigations) | 3 | 0 | 3 | 0 | 3
Weight increased (Investigations) | 2 | 0 | 2 | 0 | 2
Blood glucose increased (Investigations) | 1 | 1 | 1 | 1 | 2
Blood lactate dehydrogenase (LDH) increased (Investigations) | 1 | 1 | 1 | 1 | 2
Blood thyroid stimulating hormone (TSH) increased (Investigations) | 1 | 3 | 3 | 1 | 4
Blood urea increased (Investigations) | 1 | 1 | 1 | 1 | 2
Hepatic enzyme increased (Investigations) | 1 | 2 | 3 | 0 | 3
Electrocardiogram (ECG) ST-segment abnormal (Investigations) | 0 | 2 | 1 | 1 | 2
ECG T-wave abnormal (Investigations) | 0 | 2 | 1 | 1 | 2
Fatigue (General disorders) | 7 | 4 | 11 | 1 | 11
Peripheral edema (General disorders) | 5 | 1 | 6 | 0 | 6
Chills (General disorders) | 4 | 0 | 4 | 0 | 4
Catheter site pain (General disorders) | 2 | 0 | 2 | 0 | 2
Non-cardiac chest pain (General disorders) | 2 | 2 | 2 | 2 | 4
Pyrexia (General disorders) | 2 | 0 | 2 | 0 | 2
Pain (General disorders) | 1 | 1 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 7 | 2 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 4 | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5 | 2 | 7
Costcochondritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 1 | 4
Clubbing (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 0 | 3
Dizziness (Nervous system disorders) | 6 | 2 | 7 | 1 | 8
Headache (Nervous system disorders) | 4 | 1 | 4 | 1 | 5
Memory impairment (Nervous system disorders) | 4 | 0 | 4 | 0 | 4
Hypoesthesia (Nervous system disorders) | 2 | 0 | 2 | 0 | 2
Lethargy (Nervous system disorders) | 2 | 0 | 2 | 0 | 2
Paresthesia (Nervous system disorders) | 2 | 1 | 3 | 0 | 3
Balance disorder (Nervous system disorders) | 1 | 1 | 2 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 4 | 1 | 5 | 0 | 5
Atrial fibrillation (Cardiac disorders) | 3 | 2 | 5 | 0 | 5
Congestive cardiac failure (Cardiac disorders) | 3 | 1 | 4 | 0 | 4
Coronary artery disease (Cardiac disorders) | 2 | 2 | 4 | 1 | 4
Acute myocardial infarction (AMI) (Cardiac disorders) | 1 | 2 | 2 | 1 | 3
Angina pectoris (Cardiac disorders) | 1 | 1 | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 1 | 4 | 1 | 5
Stress fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 2
Head injuries (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1 | 2
Joint injury (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | 2
Anxiety (Psychiatric disorders) | 6 | 1 | 7 | 0 | 7
Insomnia (Psychiatric disorders) | 4 | 1 | 5 | 0 | 5
Depression (Psychiatric disorders) | 3 | 0 | 3 | 0 | 3
Panic attack (Psychiatric disorders) | 1 | 1 | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0 | 5 | 0 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0 | 3 | 0 | 3
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3 | 0 | 3
Hypertension (Vascular disorders) | 2 | 0 | 2 | 0 | 2
Hypotension (Vascular disorders) | 2 | 1 | 3 | 0 | 3
Hematuria (Renal and urinary disorders) | 1 | 1 | 1 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 2 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 2 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 2 | 0 | 2
Vision blurred (Eye disorders) | 2 | 0 | 2 | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 1 | 2 | 0 | 2
Small intestinal obstruction (General disorders) | 1 | 1 | 2 | 0 | 2
Syncope (Nervous system disorders) | 1 | 1 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/47/NCT02688647/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT02688647/SAP_001.pdf